CLINICAL TRIAL: NCT06523829
Title: The Effect of Video-Based Education on Activities of Daily Living, Wound Healing and Prosthesis Dislocation of Patients With Total Hip Replacement
Brief Title: Effect of Video Education on Daily Life Quality and Wound Care in Total Hip Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, AYŞE SİNEM TAŞ, Assistant Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BandirmaOnyediEylulU-AST-01
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Daily life activities; Wound Heal; Replacement, Hip

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled trial.
Who Masked: Participant, Care Provider
Masking Description: Participants were not informed of which group they were in when they agreed to participate in the study. Similarly, caregivers and hospital staff were not informed about the groups. Only the researcher knew which group the participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group given video-based training (Active Comparator): The application of the study to the active group;
  * In addition to routine nursing care in the ward, video and education booklet were used. Video education was given to the patient and caregiver individually in the patient room. Watching the video takes 12 minutes.
  * Video-based education was given in the preoperative period, on the 2nd-3rd postoperative day and at the discharge stage.
  Interventions: Other: GROUP GIVEN VIDEO TRAINING
- GROUP RECEIVING ROUTINE NURSING CARE (No Intervention): The application of the study to the control group; The patient was informed about the process before and after the surgery by the physician and the nurse working in the ward that day. The patient's pre-operative, surgical preparation, post-operative and discharge periods were carried out by different nurses due to work schedules. The patients were prepared by the nurse working in the ward that day on the day of surgery and sent to the operating room. After the surgery, the patients were given patient care in the ward and their follow-up and treatments were performed. During the discharge period, discharge information was given and discharge procedures were carried out.

INTERVENTIONS:
Other: GROUP GIVEN VIDEO TRAINING — Video-based training was given to this group.
  Arms: Group given video-based training

SUMMARY:
This study was conducted to examine the effects of video-based education on the activities of daily living, wound healing and prosthesis dislocation of patients who had total hip replacement surgery.

The main questions it aims to answer are:

Total hip replacement patients who received video-based education had higher postoperative daily living activities scale mean scores than patients who did not receive education.

Total hip replacement patients who received video-based education had lower postoperative Oxford Hip Score scale mean scores than patients who did not receive education.

Total hip replacement patients who received video-based education had lower postoperative Patient and Observer Scar Assessment scale mean scores than patients who did not receive education.

DETAILED DESCRIPTION:
The study was conducted in Balikesir Bandırma Education and Research Hospital, Orthopedics Clinic. Patients who met the inclusion criteria were randomly assigned to the intervention (video-based education) and control (standard nursing care) groups using randomizer.org. In collecting the study data; Individual Identification Form, Standardized Mini Mental Test, Barthel Daily Living Activities Index, Oxford Hip Score, Patient and Observer Scar Assessment Scale were used. Individual Identification Form, Barthel Daily Living Activities Index and Oxford Hip Score were applied to both groups before surgery. The intervention group received video-based education before surgery, the control group did not receive any education and received routine nursing care. On the 5th day after surgery, both groups were applied Barthel Daily Living Activities and Patient and Observer Scar Assessment Scale. Video-based education was repeated on the 2nd or 3rd day after surgery to the intervention group, and the control group received routine nursing care. Before discharge, video-based education was uploaded to the phones or computers of the patients and caregivers in the intervention group, and patients and caregivers were able to benefit from this education video whenever they wanted. Patients in the control group were discharged after receiving routine discharge education. Barthel Daily Living Activities, Oxford Hip Score and Patient and Observer Scar Assessment Scale were applied to both groups on the 30th day after surgery. Descriptive statistical methods (frequency, mean) were applied in the analysis of the data. Student t test was used in the analysis of normally distributed variables in independent groups, and the relationship between multiple independent variables was evaluated with the ANOVA test. Variance analysis was used in repeated measurements in the evaluation of quantitative data within the group. Pearson correlation analysis was used in the evaluation of the relationship between quantitative variables, and Fisher's Exact and Pearson Chi-square tests were used in the comparison of qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the study,
* Are conscious, oriented and cooperative,
* Are over 18 years of age,
* Speak Turkish,
* Are at least primary school graduates,
* Have received the Standardized Mini Mental Test and scored over 23 points according to the guideline were included.

Exclusion Criteria:

* Patients with communication problems (hearing, visual impairment)
* Patients diagnosed with a psychiatric disease
* Patients whose mobilization was not permitted by the physician were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Number of patients whose daily living activities increased thanks to video training | Change measurements for each participant were made at baseline, day 5, and day 30 after surgery.
  Barthel Daily Living Activities Index will be used to evaluate this result. Cronbach alpha value was calculated as 0.90. ADL is the most preferred evaluation index among similar indexes that evaluates the level of independence of individuals in their daily activities. Barthel Index evaluates 10 areas including nutrition, washing, dressing, self-care, bowel care, bladder care, toilet use, mobility, going up and down stairs and transferring from wheelchair to bed and the lowest score is 0 and the highest score is 100. 0-20 points indicate that the individual is fully dependent, 21-61 points indicate that the individual is highly dependent, 62-90 points indicate that the individual is moderately dependent, 91-99 points indicate that the individual is slightly dependent and 100 points indicate that the individual is fully independent. In this study, Cronbach alpha coefficient of "Barthel Daily Living Activities Index" was found as 0.859.

SECONDARY OUTCOMES:
Number of patients whose wound healing improved thanks to video training | Change measurements for each participant were made on day 5 and day 30 after surgery.
  The Patient and Observer Scar Assessment Scale (PASS) will be used to assess the wound site. The scale used to assess the wound site consists of a total of 7 items; 6 items assessing the wound in terms of flexibility, pain, color, pruritus, irregularity, and thickness, and 1 item assessing it in general. Each item has a Likert-type scoring between 1 and 10. 1 indicates "normal skin" and 10 indicates "worst scar assessment". Cronbach's alpha value of the scale was found to be 0.992 for HSDS and 0.993 for GSDÖ. In this study, Cronbach's alpha coefficient for HSDS was found to be 0.908, and for GSDÖ, Cronbach's alpha coefficient was found to be 0.953.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE SİNEM TAŞ, PHD, Principal Investigator — BANDIRMA ONYEDİ EYLÜL ÜNİVERSİTESİ
Locations (1):
- Bandirma Eğitim Ve Araştirma Hastanesi, Balıkesir, Balikesi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tas AS, Eser I. The Effect of Video-Based Education on Activities of Daily Living and Wound Healing of Patients with Total Hip Replacement: Randomised Controlled Trials. Nurs Rep. 2025 Oct 4;15(10):356. doi: 10.3390/nursrep15100356. PMID 41149671